CLINICAL TRIAL: NCT00975715
Title: A Multicentre, Randomized, Double-blind, Placebo Controlled, Parallel-group Study in Children With Inadequately Controlled Partial Onset Seizures to Investigate Efficacy, Safety and Tolerability of TRI476 (Oxcarbazepine) as Adjunctive Therapy
Brief Title: Efficacy, Safety and Tolerability of TRI476 (Oxcarbazepine) in Children With Inadequately Controlled Partial Onset Seizures
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTRI476B1301
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Results first posted 2014-01-24 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Partial Onset Seizures
Keywords: Seizures; oxcarbazepine; child
MeSH Terms: conditions — Seizures | interventions — Benzodiazepines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- TRI476 (Experimental): Participants received TRI476 based on body weight with titration up to the maintenance dose, in addition to their traditional antiepileptics dosage.
  Interventions: Drug: TRI476; Drug: Benzodiazepines
- Placebo (Placebo Comparator): Participants received placebo to TRI476 without any adjustment to the dosing regimen, in addition to their traditional antiepileptics dosage.
  Interventions: Drug: Placebo to TRI476; Drug: Benzodiazepines

INTERVENTIONS:
Drug: TRI476 — TRI476 oral suspension doses, based on body weight twice daily
  Arms: TRI476
Drug: Placebo to TRI476 — Placebo oral suspension, taken twice daily
  Arms: Placebo
Drug: Benzodiazepines — Benzodiazepines could be used as needed as rescue medication during the duration of the study.

SUMMARY:
This study is designed to provide short term efficacy and safety data of TRI476 in children with inadequately-controlled partial seizures. Patients will be randomized into either drug treatment or placebo group at 1:1 ratio, and receive their respective treatment for 8 weeks. The purpose of study is to confirm that TRI476 as adjunctive therapy is effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients, aged 4 to 14 years (inclusive), with a minimum body weight of 15 kg.
* A diagnosis of partial onset seizures, which include the seizure subtypes of simple, complex, and secondarily generalized seizures (based on the International League Against Epilepsy (ILAE) Classification, as modified in 1981).

Exclusion Criteria:

* A document history of generalized status epileptics in the past 6 months.
* Seizures having a metabolic, neoplastic, or active infectious origin.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Actual)
Dates: Start 2009-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Japan (25):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Ohbu, Aichi-ken
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Gifu, Gifu
  - Novartis Investigative Site, Kameda-gun, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kōshi, Kumamoto
  - Novartis Investigative Site, Kashiwazaki, Niigata
  - Novartis Investigative Site, Niigata, Niigata
  - Novartis Investigative Site, Yufu, Oita Prefecture
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Neyagawa, Osaka
  - Novartis Investigative Site, Higashimatsuyama-shi, Saitama
  - Novartis Investigative Site, Saitama, Saitama
  - Novartis Investigative Site, Moriyama-shi, Shiga
  - Novartis Investigative Site, Shizuoka, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Yamagata, Yamagata
  - Novartis Investigative Site, Chūō, Yamanashi

REFERENCES:
- See also: Click here for more information about this study: — http://www.novartisclinicaltrials.com/webapp/etrials/home.do

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 99 patients were randomized, one patient who did not receive study drug was excluded. A total of 48 participants were randomized to TRI476 and 51 to placebo. 7 participants discontinued during the titration period and 3 discontinued during the maintenance period. A total of 89 participants completed the study.
Pre-assignment Details: Participants kept same dosage of their traditional antiepileptics prior to screening and throughout the study. They received TRI476 or placebo in a 1:1 ratio. TRI476 dose was increased gradually, based on body weight during the titration period (day 0- 14). The tolerated dose was given during the maintenance period (up to day 56).
Period: Titration Period
Arm/Group | TRI476 | Placebo
Started | 48 | 51
Completed | 41 | 51
Not Completed | 7 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Protocol Violation | 1 | 0
Period: Maintenance Period
Arm/Group | TRI476 | Placebo
Started | 41 | 51
Completed | 39 | 50
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRI476 | Placebo | Total
Number analyzed (Participants) | 48 | 51 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (2.91) | 9.2 (2.83) | 9.5 (2.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 26 | 27 | 53

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Partial Onset Seizure Frequency Per 28 Days From Baseline to the Double-blind Phase, by Treatment Group
Description: Percent change in partial onset seizure frequency per 28 days during the double-blind phase from the screening phase, was calculated according to the following formula: "Percent change in partial onset seizure frequency per 28 days from the screening phase" = (partial onset seizure frequency per 28 days during the double-blind phase - partial onset seizure frequency per 28 days during the screening phase) / partial onset seizure frequency per 28 days during the double-blind phase x 100 "Partial onset seizure frequency per 28 days" = Number of partial onset seizures during each phase (screening phase or double-blind phase) / number of days during the screening or double-blind phase × 28.
Time Frame: screening and 28 days
Population: The Full Analysis set included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: percentage change per 28 days
Arm/Group | TRI476 | Placebo
Number analyzed (Participants) | 47 | 51
percentage change per 28 days | -2.85 (63.546) | 14.82 (73.333)

2. Secondary Outcome: Partial Seizure Frequency Per 28 Days, by Study Period (Every 28 Days) and Treatment Group
Description: Partial onset seizure frequency per 28 days during a period between baseline and Week 4 was measured. Partial onset seizure frequency per 28 days (count/28 days)" = Number of partial onset seizures during each phase (screening phase or double-blind phase) / Number of days during the phase x 28.
Time Frame: baseline, 28 days and 56 days
Population: The Full Analysis set included all participants who received study drug.
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Arm/Group | TRI476 | Placebo
Number analyzed (Participants) | 47 | 51
seizures per 28 days
  Baseline to Week 4 (day 0 to day 28) | 65.58 (109.457) | 90.61 (283.187)
  Week 4 to Week 8 (day 28 to day 56) | 45.40 (70.209) | 98.73 (291.781)

3. Secondary Outcome: Percent of Participants With Response During Double-blind Phase, by Treatment Group
Description: Responder rate was defined as the percent of participants with an at least 50% reduction in partial onset seizure frequency per 28 days from the screening phase.
Time Frame: screening to 28 days
Population: The Full Analysis set included all participants who received study drug.
Measure: Number; unit: percentage of participants
Arm/Group | TRI476 | Placebo
Number analyzed (Participants) | 47 | 51
percentage of participants | 23.4 | 3.9

4. Secondary Outcome: Percent Change in Partial Onset Seizure Frequency During the Double-blind Phase by Seizure Type
Description: Percent change in seizure frequency from baseline = 100 (T-B)/B, B=Seizure frequency per 28 days during baseline phase, T=Seizure frequency per 28 days during the double-blind phase. Seizure frequency per 28 days is calculated as: (seizure frequency during the double-blind phase / the number of days the seizure information were provided) x 28. Only patients with both baseline and corresponding post-baseline values are included.
Time Frame: 28 days
Population: Analyzed set includes all participants who received study drug and had both baseline and post baseline data available.
Measure: Mean (Standard Deviation); unit: percentage change in seizure frequency
Arm/Group | TRI476 | Placebo
Number analyzed (Participants) | 47 | 51
percentage change in seizure frequency
  Simple partial seizures | -9.73 (51.329) | -16.89 (45.822)
  Complex partial seizures | -6.86 (78.583) | 30.59 (91.551)
  Secondarily generalized seizures | -29.54 (64.660) | 12.11 (82.879)

5. Secondary Outcome: Number of Participants With Clinical Global Impression of Change (CGIC) at Final Assessment, by Treatment Group
Description: Clinical Global Impression of Change (CGI) is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients). CGI-C scores range from 1 (very much improved) through to 7 (very much worse).
Time Frame: 56 days
Population: The Analysis set included all participants who received study drug and had data available for analysis.
Measure: Number; unit: participants
Arm/Group | TRI476 | Placebo
Number analyzed (Participants) | 47 | 51
participants
  Marked improvement | 9 | 2
  Moderate improvement | 8 | 2
  Slight improvement | 8 | 6
  No change | 21 | 38
  Slight aggravation | 1 | 3
  Moderate aggravation | 0 | 0
  Marked aggravation | 0 | 0

ADVERSE EVENTS:
Description: A total of 99 patients were randomized, one patient who did not receive study drug was excluded from the safety analysis set
Arm/Group | TRI476 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/47 | 1/51
Other Adverse Events (participants affected / at risk) | 38/47 | 27/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRI476 (N=47) | Placebo (N=51)
Bronchopneumonia (Infections and infestations) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TRI476 (N=47) | Placebo (N=51)
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Conjunctivitis (Eye disorders) | 2 | 2
Diplopia (Eye disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 5 | 3
Pyrexia (General disorders) | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 5 | 9
Otitis media (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Contusion (Injury, poisoning and procedural complications) | 2 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Ataxia (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 20 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.